CLINICAL TRIAL: NCT04740827
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-controlled, Parallel-Group Study to Evaluate the Efficacy, Safety, and Tolerability of Oral Atogepant for the Prophylaxis of Migraine in Participants With Episodic Migraine Who Have Previously Failed 2 to 4 Classes of Oral Prophylactic Treatments (ELEVATE)
Brief Title: Atogepant for Prophylaxis of Migraine in Participants Who Failed Previous Oral Prophylactic Treatments.
Acronym: ELEVATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3101-304-002; 2019-003448-58 (EudraCT Number)
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Episodic Migraine
Keywords: Episodic migraine
MeSH Terms: interventions — atogepant

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received atogepant-matching placebo tablets, orally, once daily (QD) for up to 12 weeks in a double-blind (DB) treatment period.
  Interventions: Drug: Placebo
- Atogepant 60 mg (Active Comparator): Participants received atogepant 60 mg, orally, QD for up to 12 weeks in a DB treatment period.
  Interventions: Drug: Atogepant 60 mg

INTERVENTIONS:
Drug: Atogepant 60 mg — Atogepant tablets.
  Arms: Atogepant 60 mg
Drug: Placebo — Atogepant matching placebo tablets.
  Arms: Placebo

SUMMARY:
This study will assess the safety, tolerability, and efficacy of Atogepant 60 mg compared with placebo in participants with episodic migraine and who have previously failed 2 to 4 classes of oral prophylactic treatments.

ELIGIBILITY:
Inclusion Criteria:

* At least a 1-year history of migraine with or without aura consistent with a diagnosis according to the ICHD-3, 2018.
* Age of the participant at the time of migraine onset < 50 years -History of 4 to 14 migraine days per month on average in the 3 months prior to Visit 1 in the investigator's judgment
* Female participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period. Male participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period.
* 4 to 14 migraine days in the 28-day baseline period per eDiary
* Failed oral migraine prophylaxis medications from 2 to 4 medication classes

Exclusion Criteria:

* Any clinically significant hematologic, endocrine, pulmonary, hepatic, gastrointestinal, or neurologic disease
* Participant has any other concurrent pain condition that, in the opinion of the investigator, may significantly impact the current headache disorder
* In the opinion of the investigator, confounding psychiatric conditions, dementia, epilepsy, or significant neurological disorders other than migraine
* Has ≥ 15 headache days per month on average across the 3 months prior to Visit 1 in the investigator's judgment
* Has ≥ 15 headache days in the 28-day baseline period per eDiary
* Clinically significant cardiovascular or cerebrovascular disease
* Has a history of migraine accompanied by diplopia or decreased level of consciousness or retinal migraine as defined by ICHD-3, 2018
* Has a current diagnosis of chronic migraine, new persistent daily headache, medication overuse headache, trigeminal autonomic cephalgia (eg, cluster headache), or painful cranial neuropathy as defined by ICHD-3, 2018

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (114):
- United States (26):
  - Axiom Research /ID# 226379, Colton, California
  - Pharmacology Research Institute (PRI) - Encino (Wake) /ID# 226434, Encino, California
  - Pharmacology Research Institute (PRI) - Los Alamitos (Wake) /ID# 226388, Los Alamitos, California
  - Pharmacology Research Institute (PRI) - Los Alamitos (Wake) /ID# 226405, Los Alamitos, California
  - Excell Research, Inc /ID# 228386, Oceanside, California
  - Alpine Clinical Research Center /ID# 226201, Boulder, Colorado
  - Sensible Healthcare /ID# 226197, Ocoee, Florida
  - Meridien Research /ID# 226224, St. Petersburg, Florida
  - Meridien Research /ID# 226302, St. Petersburg, Florida
  - Velocity Clinical Research - Boise /ID# 226320, Meridian, Idaho
  - Allied Physicians - Fort Wayne Neurological Center /ID# 226350, Fort Wayne, Indiana
  - Deaconess Clinic - Gateway Health Center /ID# 226481, Newburgh, Indiana
  - Pharmasite Research, Inc. /ID# 226445, Baltimore, Maryland
  - StudyMetrix Research /ID# 226297, City of Saint Peters, Missouri
  - Clinvest Research LLC /ID# 226273, Springfield, Missouri
  - Methodist Physicians Clinic /ID# 226470, Fremont, Nebraska
  - Amici Clinical Research - Raritan /ID# 226282, Raritan, New Jersey
  - Albuquerque Clinical Trials, Inc /ID# 233445, Albuquerque, New Mexico
  - CTI Clinical Trial and Consulting /ID# 226281, Cincinnati, Ohio
  - FutureSearch Trials of Neurology /ID# 226423, Austin, Texas
  - Austin Clinical Trial Partners /ID# 228387, Austin, Texas
  - DiscoveResearch, Inc /ID# 226491, Bryan, Texas
  - FutureSearch Trials of Dallas, LP /ID# 226493, Dallas, Texas
  - LinQ Research, LLC /ID# 226227, Pearland, Texas
  - Highland Clinical Research /ID# 226288, Salt Lake City, Utah
  - Northwest Clinical Research Center /ID# 226228, Bellevue, Washington
- Australia (2):
  - Alfred Health /ID# 226341, Melbourne, Victoria
  - The Royal Melbourne Hospital /ID# 226402, Parkville, Victoria
- Canada (3):
  - Aggarwal and Associates Limited /ID# 226321, Brampton, Ontario
  - Ottawa Headache Centre Research Inc /ID# 226257, Ottawa, Ontario
  - Diex Recherche Sherbrooke Inc. /ID# 226375, Sherbrooke, Quebec
- Czechia (12):
  - POLIKLINIKA CHOCEN, a.s. /ID# 226510, Choceň
  - BRAIN-SOULTHERAPY s.r.o. /ID# 226489, Kladno
  - CCR Ostrava, s.r.o. /ID# 226279, Ostrava
  - A-SHINE s.r.o. /ID# 226208, Pilsen
  - CLINTRIAL s.r.o. /ID# 226192, Prague
  - DADO MEDICAL s.r.o. /ID# 226548, Prague
  - CCR Prague s.r.o. /ID# 226214, Prague
  - CCR Czech a.s /ID# 226270, Prague
  - FORBELI s.r.o. /ID# 226396, Prague
  - INEP medical s.r.o. /ID# 226531, Prague
  - Vestra Clinics s.r.o. /ID# 226547, Rychnov nad Kněžnou
  - NeuroMed Zlin s.r.o. /ID# 226487, Zlín
- Rigshospitalet Glostrup /ID# 226271, Glostrup Municipality, Capital Region, Denmark
- France (5):
  - CHU Nice - Hopital de Cimiez /ID# 226401, Nice, Alpes-Maritimes
  - CHU Lille /ID# 226501, Lille, Nord
  - CHU de SAINT ETIENNE - Hopital Nord /ID# 226397, Saint Priest EN Jarez, Pays de la Loire Region
  - CHU Clermont Ferand - Hopital Gabriel Montpied /ID# 226438, Clermont-Ferrand
  - AP-HP - Hopital Lariboisière /ID# 226221, Paris
- Germany (17):
  - Universitaetsklinikum Tuebingen /ID# 226529, Tübingen, Baden-Wurttemberg
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 226441, Berlin
  - Klinische Forschung Dresden GmbH /ID# 226194, Dresden
  - Praxis Dr. Gendolla /ID# 226497, Essen
  - Universitaetsklinikum Essen /ID# 226527, Essen
  - Klinische Forschung Hannover-Mitte GmbH /ID# 226195, Hanover
  - Universitaetsklinikum Jena Klinik fuer Neurologie /ID# 226439, Jena
  - Vitos Orthopaedische Klinik Kassel gemeinnuetzige GmbH /ID# 231767, Kassel
  - Schmerzklinik Kiel /ID# 226499, Kiel
  - AmBeNet GmbH /ID# 226213, Leipzig
  - Pharmakologisches Studienzentrum Chemnitz GmbH /ID# 226202, Mittweida
  - Universitaetsmedizin Rostock /ID# 226517, Rostock
  - Neuropoint GmbH /ID# 226377, Ulm
  - Neuropraxis Muenchen Sued /ID# 226216, Unterhaching
  - Studienzentrum Nord-West /ID# 226360, Westerstede
  - Intermed GmbH /ID# 226376, Wiesbaden
  - DKD Helios Klinik Wiesbaden /ID# 226534, Wiesbaden
- Hungary (7):
  - Bugat Pal Korhaz /ID# 226357, Gyöngyös, Heves County
  - Valeomed Kft /ID# 226535, Esztergom, Komárom-Esztergom
  - Szent Borbala Korhaz /ID# 226400, Tatabánya, Komárom-Esztergom
  - Somogy Megyei Kaposi Mor Oktato Korhaz /ID# 226485, Kaposvár, Somogy County
  - Mind Klinika Kft. /ID# 233438, Budapest
  - Clinexpert Kft /ID# 226467, Budapest
  - Department of Neurology, University of Szeged /ID# 226442, Szeged
- Italy (7):
  - Ospedale Ss. Filippo e Nicola /ID# 226530, Avezzano, L Aquila
  - Fondazione Policlinico Universitario Campus Bio-Medico di Roma /ID# 226361, Rome, Lazio
  - Univ. of Bologna-IRCCS-Istituto delle Scienze Neurologiche /ID# 226475, Bologna
  - Azienda Ospedaliero Universitaria Careggi /ID# 226502, Florence
  - Fondazione IRCCS Istituto Neurologico Carlo Besta /ID# 226399, Milan
  - AOU Universita degli Studi della Campania Luigi Vanvitelli /ID# 226503, Napoli
  - Universita di Pavia /ID# 226536, Pavia
- Netherlands (3):
  - Martini Ziekenhuis /ID# 226343, Groningen
  - Canisius-Wilhelmina Ziekenhuis /ID# 226488, Nijmegen
  - ZorgSaam Zorggroep Zeeuws-Vlaanderen /ID# 226317, Terneuzen
- Poland (11):
  - Solumed Centrum Medyczne /ID# 226299, Poznan, Greater Poland Voivodeship
  - NZOZ Vitamed /ID# 226293, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczne Gabinety Sp. z o.o. /ID# 226266, Krakow, Lesser Poland Voivodeship
  - Centrum Leczenia Padaczki i Migreny /ID# 226543, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Oporow /ID# 226469, Wroclaw, Lower Silesian Voivodeship
  - Indywidualna Praktyka Lekarska dr hab. med. Anna Szczepanska-Szerej /ID# 226235, Lublin, Lublin Voivodeship
  - Duplicate_RCMed Oddzial Sochaczew /ID# 226369, Sochaczew, Masovian Voivodeship
  - Centrum Medyczne Pratia Gdynia /ID# 226437, Gdynia, Pomeranian Voivodeship
  - Silmedic Sp. z o.o. /ID# 226267, Katowice, Silesian Voivodeship
  - EuroMedis sp. z o.o. /ID# 226268, Szczecin, West Pomeranian Voivodeship
  - Gabinet Lekarski Jacek Rozniecki /ID# 226323, Lodz, Łódź Voivodeship
- Russia (5):
  - Bashkir State Medical University /ID# 226552, Ufa, Bashkortostan Republic
  - Kazan State Medical University /ID# 226498, Kazan', Tatarstan, Respublika
  - Sbhi Cp 2 Hdm /Id# 226494, Moscow
  - University Headache Clinic /ID# 226435, Moscow
  - Cephalgolog /ID# 226541, Moscow
- Spain (7):
  - Hospital Unversitario Marques de Valdecilla /ID# 226239, Santander, Cantabria
  - University Clinical Hospital of Valladolid /ID# 226528, Valledolid, Castellon
  - Hospital Universitario Vall d'Hebron /ID# 226230, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 226550, Barcelona
  - Hospital Clinico Universitario San Carlos /ID# 226483, Madrid
  - Hospital Clinico Universitario de Valencia /ID# 226472, Valencia
  - Hospital Clinico Universitario Lozano Blesa /ID# 226395, Zaragoza
- Karolinska university hospital, Huddinge /ID# 226215, Huddinge, Stockholm County, Sweden
- United Kingdom (7):
  - Queen Elizabeth University Hospital /ID# 226492, Glasgow
  - Re:Cognition Health - Guildford /ID# 226539, Guildford
  - NHS Highland /ID# 226542, Inverness
  - Leeds Teaching Hospitals NHS Trust /ID# 226538, Leeds
  - St Pancras Clinical Research /ID# 226551, London
  - King's College Hospital NHS Foundation Trust /ID# 226525, London
  - Re:Cognition Health - London /ID# 226540, London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Goadsby PJ, Jurgens TP, Brand-Schieber E, Nagy K, Liu Y, Boinpally R, Stodtmann S, Trugman JM. Efficacy of ubrogepant and atogepant in males and females with migraine: A secondary analysis of randomized clinical trials. Cephalalgia. 2025 Feb;45(2):3331024251320610. doi: 10.1177/03331024251320610. PMID 39982105
- [Derived] Lipton RB, Gandhi P, Tassorelli C, Reuter U, Harriott AM, Holle-Lee D, Gottschalk CH, Neel B, Liu Y, Guo H, Stokes J, Nagy K, Dabruzzo B, Smith JH. Early Improvements With Atogepant for the Preventive Treatment of Migraine: Results From 3 Randomized Phase 3 Trials. Neurology. 2025 Jan 28;104(2):e210212. doi: 10.1212/WNL.0000000000210212. Epub 2024 Dec 23. PMID 39715475
- [Derived] Gottschalk C, Gandhi P, Pozo-Rosich P, Christie S, Tassorelli C, Stokes J, Liu Y, Luo L, Nagy K, Trugman JM, Lipton RB. Effect of preventive treatment with atogepant on quality of life, daily functioning, and headache impact across the spectrum of migraine: Findings from three double-blind, randomized, phase 3 trials. Cephalalgia. 2024 Dec;44(12):3331024241300305. doi: 10.1177/03331024241300305. PMID 39648617
- [Derived] Tassorelli C, Nagy K, Pozo-Rosich P, Lanteri-Minet M, Sacco S, Nezadal T, Guo H, De Abreu Ferreira R, Forero G, Trugman JM. Safety and efficacy of atogepant for the preventive treatment of episodic migraine in adults for whom conventional oral preventive treatments have failed (ELEVATE): a randomised, placebo-controlled, phase 3b trial. Lancet Neurol. 2024 Apr;23(4):382-392. doi: 10.1016/S1474-4422(24)00025-5. Epub 2024 Feb 13. PMID 38364831

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 315 participants were randomized to receive atogepant-matching placebo or atogepant in a double-blind treatment period, and 313 participants received at least 1 dose of study intervention (safety population). From the 295 participants who completed the double-blind period 87 participants entered the follow-up period. Participants who rolled over directly at Week 12 to study 3101-312-002 [NCT04686136] did not enter the safety-follow up period.
Period: Double-blind Treatment (Up to Week 12)
Arm/Group | Placebo | Atogepant 60 mg
Started | 158 | 157
Safety Population (Safety population consisted of all participants who received at least 1 dose of study intervention.) | 157 | 156
Modified Intent-to-Treat (mITT) Population (mITT population consisted of all randomized participants who received at least 1 dose of study intervention, had an evaluable baseline period of eDiary data, and had at least 1 evaluable postbaseline 4-week period (Weeks 1 to 4, 5 to 8, and 9 to 12) of eDiary data during the double-blind treatment period.) | 154 | 151
Off-treatment Hypothetical Estimand (OTHE) Population (OTHE population consisted of all randomized participants who received at least 1 dose of study intervention, had an evaluable baseline period of eDiary data, and had at least 1 evaluable postbaseline 4-week period (Weeks 1 to 4, 5 to 8, 9 to 12) of eDiary data, regardless of whether on study intervention or off study intervention.) | 155 | 154
Completed | 151 | 144
Not Completed | 7 | 13
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Deviation | 3 | 5
Period: Follow-up Period (Week 13 to Week 16)
Arm/Group | Placebo | Atogepant 60 mg
Started (Of 295 participants who completed the double-blind period 87 participants entered the follow-up period. Participants who rolled over directly at Week 12 to study 3101-312-002 [NCT04686136] did not enter the safety-follow up period.) | 43 | 44
Completed | 42 | 44
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all randomized participants.
Groups:
- Placebo: Participants received atogepant-matching placebo tablets, orally, QD for up to 12 weeks in a DB treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Atogepant 60 mg | Total
Number analyzed (Participants) | 158 | 157 | 315
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (10.29) | 40.8 (10.71) | 42.1 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 140 | 281
  Male | 17 | 17 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 154 | 150 | 304
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 152 | 150 | 302
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Monthly Migraine Days in mITT Population [Mean (Standard Deviation); unit: Migraine days per month] — A migraine day was any calendar day on which the participant experienced a migraine headache. The monthly (4-week) migraine days was defined as the total number of reported migraine days in diary divided by total number of days with diary records during each 4-week period and multiplied by 28. Population: mITT population included all randomized participants who received at least 1 dose of study intervention.
  Migraine days per month
    number analyzed (Participants) | 154 | 151 | 305
    (all) | 9.3 (2.41) | 9.0 (2.30) | 9.2 (2.35)
Monthly Migraine Days in OTHE Population [Mean (Standard Deviation); unit: Migraine days per month] — A migraine day was any calendar day on which the participant experienced a migraine headache. The monthly (4-week) migraine days was defined as the total number of reported migraine days in diary divided by total number of days with diary records during each 4-week period and multiplied by 28. Population: OTHE population consisted of all randomized participants who received at least 1 dose of study intervention, had an evaluable baseline period of eDiary data, and had at least 1 evaluable postbaseline 4-week period (Weeks 1 to 4, 5 to 8, 9 to 12) of eDiary data, regardless of whether on study intervention or off study intervention.
  Migraine days per month
    number analyzed (Participants) | 155 | 154 | 309
    (all) | 9.3 (2.40) | 9.1 (2.29) | 9.2 (2.34)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Monthly Migraine Days Across 12-Week Treatment Period in mITT Population
Description: Participants recorded daily duration of migraine in a diary. A migraine day was any calendar day on which the participant experienced a migraine headache. The monthly (4-week) migraine days were defined as the total number of reported migraine days in diary divided by total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Baseline is defined as the number of migraine days during the last 28 days prior to the randomization date. Negative change from Baseline indicates improvement. Mixed-effects model for repeated measures (MMRM) was used for analysis.
Time Frame: Baseline to Week 12
Population: mITT Population included all randomized participants who received at least 1 dose of study treatment, had an evaluable baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period of eDiary data during the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: migraine days per month
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 154 | 151
migraine days per month | -1.86 (0.389) | -4.29 (0.397)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < 0.0001, MMRM; Least Squares Mean Difference = -2.43, 95% CI 2-sided [-3.27 to -1.59], Standard Error of Mean 0.426 — MMRM=baseline monthly migraine days as covariate, treatment group, visit, region and number of classes of failed prior treatments as fixed factors; treatment group and baseline-by-visit as interaction terms, with an unstructured covariance matrix

2. Primary Outcome: Change From Baseline in Mean Monthly Migraine Days Across 12-Week Treatment Period in OTHE Population
Description: Participants recorded daily duration of migraine in a diary. A migraine day was any calendar day on which the participant experienced a migraine headache. The monthly (4-week) migraine days were defined as the total number of reported migraine days in diary divided by total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Baseline is defined as the number of migraine days during the last 28 days prior to the randomization date. Negative change from Baseline indicates improvement. MMRM was used for analysis.
Time Frame: Baseline to Week 12
Population: OTHE Population included all randomized participants who received at least 1 dose of study treatment, had an evaluable baseline period of eDiary data and had at least 1 evaluable post-baseline 4-week period (Weeks 1 to 4, 5 to 8, 9 to 12) of eDiary data, regardless of whether on study treatment or off study treatment.
Measure: Least Squares Mean (Standard Error); unit: migraine days per month
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 155 | 154
migraine days per month | -1.85 (0.388) | -4.20 (0.393)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < 0.0001, MMRM; Least Squares Mean Difference = -2.35, 95% CI 2-sided [-3.19 to -1.52], Standard Error of Mean 0.425 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With At Least a 50% Reduction in 3-Month Average of Monthly Migraine Days Across the 12-week Treatment Period in mITT Population
Description: Data is reported for 50% responders averaged at each 4-week period. 50% responders are participants with at least a 50% reduction from baseline in 3-month average of monthly migraine days. Participants recorded daily duration of migraine in a diary. A migraine day was any calendar day on which the participant experienced a migraine headache. The monthly (4-week) migraine days are equal to total number of reported migraine days in diary divided by total number of days with diary records in each 4-week period multiplied by 28.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 154 | 151
Participants | 27 | 77
Statistical Analysis 1: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 5.15, 95% CI 2-sided [3.02 to 8.79] — Odds ratio and p-value are based on logistic regression with treatment group, region, baseline monthly migraine days, and number of classes of failed prior prophylactic treatments (2 and >2) as explanatory variables

4. Secondary Outcome: Number of Participants With At Least a 50% Reduction in 3-Month Average of Monthly Migraine Days Across the 12-week Treatment Period in OTHE Population
Description: as for outcome 3
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 155 | 154
Participants | 28 | 78
Statistical Analysis 1: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.82, 95% CI 2-sided [2.85 to 8.14] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline in Mean Monthly Headache Days Across the 12-week Treatment Period in mITT Population
Description: Participants recorded daily total duration of a headache in a diary. A headache day is any calendar day on which the participant experienced a headache pain lasting 2 hours or longer unless an acute headache medication was used after the start of the headache. The monthly (4-week) headache days were defined as the total number of reported headache days in the diary divided by the total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Baseline is defined as the number of headache days during the last 28 days prior to the randomization date. Negative change from Baseline indicates improvement. MMRM was used for analysis.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: headache days per month
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 154 | 151
headache days per month | -1.93 (0.424) | -4.21 (0.431)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < 0.0001, MMRM; Least Squares Mean Difference = -2.28, 95% CI 2-sided [-3.15 to -1.42], Standard Error of Mean 0.440 — MMRM=baseline as covariate, treatment group, visit, region, number of classes of failed prior treatments, number of migraine days during baseline period as fixed factors; treatment group and baseline-by-visit with an unstructured covariance matrix

6. Secondary Outcome: Change From Baseline in Mean Monthly Headache Days Across the 12-week Treatment Period in OTHE Population
Description: as for outcome 5
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: headache days per month
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 155 | 154
headache days per month | -1.91 (0.423) | -4.10 (0.429)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < 0.0001, MMRM; Least Squares Mean Difference = -2.19, 95% CI 2-sided [-3.05 to -1.32], Standard Error of Mean 0.439 — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Change From Baseline in Mean Monthly Acute Medication Use Days Across the 12-week Treatment Period in mITT Population
Description: An acute medication use day is defined as any day on which a participant reports, per eDiary, the intake of allowed medication(s) to treat an acute migraine. The monthly (4-week) acute medication use days were defined as the total number of reported acute medication use days in the diary divided by the total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Baseline is defined as the number of migraine days during the last 28 days prior to the randomization date. A negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: acute medication use days per month
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 154 | 151
acute medication use days per month | -1.11 (0.359) | -3.79 (0.363)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < 0.0001, MMRM; Least Squares Mean Difference = -2.68, 95% CI 2-sided [-3.43 to -1.93], Standard Error of Mean 0.381 — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Change From Baseline in Mean Monthly Acute Medication Use Days Across the 12-week Treatment Period in OTHE Population
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: acute medication use days per month
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 155 | 154
acute medication use days per month | -1.10 (0.358) | -3.70 (0.361)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < 0.0001, MMRM; Least Squares Mean Difference = -2.61, 95% CI 2-sided [-3.36 to -1.86], Standard Error of Mean 0.380 — [estimate comment as in outcome 5, analysis 1]

9. Secondary Outcome: Change From Baseline in Migraine Specific Quality of Life Questionnaire (MSQ) v2.1 Role Function-Restrictive Domain Score at Week 12 in mITT Population
Description: The MSQ v2.1 is a 14-item questionnaire designed to measure health-related quality of life impairments attributed to migraine in the past 4 weeks. It is divided into 3 domains: Role Function Restrictive (question numbers 1-7, score ranges 7 to 42) assesses how migraines limit one's daily social and work-related activities; Role Function Preventive (question numbers 8-11, score ranges 4 to 24) assesses how migraines prevent these activities; and the Emotional Function (question numbers 12-14, score ranges 3 to 18) domain assesses the emotions associated with migraines. Participants respond to items using a 6-point scale ranging from none of the time to all of the time. Raw dimension scores are computed as a sum of item responses and rescaled to a 0 to 100 scale, where higher scores indicate better quality of life. MMRM was used for analysis.
Time Frame: Baseline to Week 12
Population: mITT Population included all randomized participants who received at least 1 dose of study treatment, had an evaluable baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period of eDiary data during the double-blind treatment period. Overall number of participants analyzed are the number of participants available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 149 | 144
score on a scale | 15.41 (2.078) | 33.09 (2.102)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < 0.0001, MMRM; Least Squares Mean Difference = 17.67, 95% CI 2-sided [13.05 to 22.30], Standard Error of Mean 2.348 — [estimate comment as in outcome 5, analysis 1]

10. Secondary Outcome: Change From Baseline in Migraine Specific Quality of Life Questionnaire (MSQ) v2.1 Role Function-Restrictive Domain Score at Week 12 in OTHE Population
Description: as for outcome 9
Time Frame: Baseline to Week 12
Population: OTHE Population included all randomized participants who received at least 1 dose of study treatment, had an evaluable baseline period of eDiary data and had at least 1 evaluable post-baseline 4-week period (Weeks 1 to 4, 5 to 8, 9 to 12) of eDiary data, regardless of whether on study treatment or off study treatment. Overall number of participants analyzed is the number of participants available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 148 | 144
score on a scale | 15.38 (2.047) | 33.26 (2.065)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < 0.0001, MMRM; Least Squares Mean Difference = 17.88, 95% CI 2-sided [13.34 to 22.42], Standard Error of Mean 2.308 — [estimate comment as in outcome 5, analysis 1]

11. Secondary Outcome: Change From Baseline in Mean Monthly Performance of Daily Activities Domain Score of the Activity Impairment in Migraine - Diary (AIM-D) Across the 12-Week Treatment Period in mITT Population
Description: The AIM-D is a 11-item patient-reported outcome (PRO) measure that assesses the impact of migraine on the performance of daily activities which include, 7 items: difficulty with household chores, errands, leisure activities at home, leisure or social activities outside the home, strenuous physical activities, concentrating, and thinking clearly and physical impairment; 4 items: difficulty walking, moving body, bending forward, moving head using a 6-point rating scale where 0=not difficult at all, 1=a little difficult, 2=somewhat difficult, 3=very difficult, 4=extremely difficult, and 5=I could not do it at all. The raw performance of daily activities domain scores were transformed to 0-100 scale, with higher scores indicating greater impact of migraine (higher disease burden).
Time Frame: Baseline to Week 12
Population: mITT Population included all randomized participants who received at least 1 dose of study treatment, had an evaluable baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period of eDiary data during the double-blind treatment period. Overall number of participants analyzed is the number of participants available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 150 | 145
score on a scale | -4.97 (0.800) | -9.68 (0.826)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < 0.0001, MMRM; Least Squares Mean Difference = -4.71, 95% CI 2-sided [-6.37 to -3.05], Standard Error of Mean 0.844 — [estimate comment as in outcome 5, analysis 1]

12. Secondary Outcome: Change From Baseline in Mean Monthly Physical Impairment Domain Score of the AIM-D Across the 12-Week Treatment Period in mITT Population
Description: The AIM-D is a 11-item PRO measure that assesses the impact of migraine on the performance of daily activities which includes 7 items: difficulty with household chores, errands, leisure activities at home, leisure or social activities outside the home, strenuous physical activities, concentrating, and thinking clearly and physical impairment; 4 items: difficulty walking, moving body, bending forward, moving head using a 6-point rating scale where 0=not difficult at all, 1=a little difficult, 2=somewhat difficult, 3=very difficult, 4=extremely difficult, and 5=I could not do it at all. The raw physical impairment domain scores were transformed to 0-100 scale, with higher scores indicating greater impact of migraine (higher disease burden).
Time Frame: Baseline to Week 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 150 | 145
score on a scale | -3.03 (0.748) | -7.43 (0.773)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < 0.0001, MMRM; Least Squares Mean Difference = -4.39, 95% CI 2-sided [-5.94 to -2.85], Standard Error of Mean 0.786 — [estimate comment as in outcome 5, analysis 1]

13. Secondary Outcome: Change From Baseline in the Headache Impact Test (HIT-6) Total Score at Week 12 in OTHE Population
Description: HIT-6 is a 6-question assessment used to measure the impact headaches have on a participant's ability to function on the job, at school, at home, and in social situations. It assesses the effect that headaches have on normal daily life and the participant's ability to function. Responses are based on frequency using a 5-point scale ranging from "never" to "always." The HIT-6 total score, which ranges from 36 to 78, is the sum of the responses - each of which is assigned a score ranging from 6 points (never) to 13 points (always). MMRM was used for the analyses.
Time Frame: Baseline to Week 12
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 148 | 144
score on a scale | -4.14 (0.795) | -10.56 (0.804)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < 0.0001, MMRM; Least Squares Mean Difference = -6.42, 95% CI 2-sided [-8.22 to -4.63], Standard Error of Mean 0.912 — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Number of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. TEAEs were defined as any AE with the onset that was after the first dose of study intervention.
Time Frame: From first dose of study drug until 30 days after last dose of study drug (up to Week 12)
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Atogepant 60 mg
Number analyzed (Participants) | 157 | 156
Participants | 84 | 81

ADVERSE EVENTS:
Time Frame: All cause mortality is reported from enrollment to end of study; median time on follow up was 93.5 and 90.0 days for Placebo and Atogepant, respectively. TEAEs and SAEs were collected from first dose of study drug until 30 days after last dose of study drug; mean duration on study drug was 83.7 days and 81.7 days for Placebo and Atogepant, respectively.
Description: All-cause mortality is reported for all participants enrolled in the study. Serious and other adverse events are reported for Safety population which consisted of all participants who received at least 1 dose of study intervention.
Arm/Group | Placebo | Atogepant 60 mg
All-Cause Mortality (participants affected / at risk) | 0/158 | 0/157
Serious Adverse Events (participants affected / at risk) | 0/157 | 4/156
Other Adverse Events (participants affected / at risk) | 34/157 | 40/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=157) | Atogepant 60 mg (N=156)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
BREAST CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INVASIVE BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ABORTION INDUCED (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=157) | Atogepant 60 mg (N=156)
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 16 (18)
NAUSEA (Gastrointestinal disorders) | 5 (5) | 11 (12)
COVID-19 (Infections and infestations) | 15 (15) | 13 (13)
NASOPHARYNGITIS (Infections and infestations) | 12 (12) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT04740827/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT04740827/SAP_001.pdf